Title: Investigating ELSI issues that may facilitate or impede clinical translation of epigenetic research: National Survey

NCT: Not yet assigned

Document Approval Date: 3/31/25



FOR IRB USE ONLY IRB ID #: 202503082 APPROVAL DATE: 03/31/25

APPROVAL DATE: 03/31/25 RELEASED DATE: 04/01/25 EXPIRATION DATE: N/A

We invite you to participate in a research study being conducted by investigators from Washington University in St. Louis. If you agree to participate in this study, you will be asked to answer survey questions and watch a brief video. The goal is to understand people's opinions about how people's genes, behaviors and environments can affect their health. The survey and video will take about 20 minutes to complete.

If you have any questions about the research study itself please contact: **Julia Maki at waterslab@wustl.edu**. If you have questions, concerns, or complaints about your rights as a research participant, please contact the Human Research Protection Office at 1-(800)-438-0445 or email <a href="mailto:hrpo@wustl.edu">hrpo@wustl.edu</a>. Thank you very much for your consideration of this research study.